CLINICAL TRIAL: NCT04944914
Title: Camrelizumab Plus Stereotactic Body Radiotherapy vs Camrelizumab Alone For Oligometastatic Nasopharyngeal Carcinoma: A Multicenter Randomized Clinical Phase 3 Trial
Brief Title: Camrelizumab Plus Stereotactic Body Radiotherapy vs Camrelizumab Alone For Oligometastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, professor & chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2021-
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Oligometastatic Nasopharyngeal Carcinoma; Immunotherapy; Stereotactic Body Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab Plus Stereotactic Body Radiotherapy (Experimental): Patients receive camrelizumab(200mg, iv drip for over 60min) every 2 weeks from 2 weeks before radiotherapy, and then receive stereotactic body radiotherapy until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, investigator decision or the upper limit of treatment duration of 1 year.
  Interventions: Drug: camrelizumab; Radiation: stereotactic body radiotherapy
- Camrelizumab (Active Comparator): Patients receive camrelizumab(200mg, iv drip for over 60min) every 2 weeks until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, investigator decision or the upper limit of treatment duration of 1 year.
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab — Patients receive camrelizumab(200mg, iv drip for over 60min) every 2 weeks from 2 weeks before radiotherapy
Radiation: stereotactic body radiotherapy — Patients receive stereotactic body radiotherapy for all oligometastatic lesions as radical therapy to control the disease and reduce any potential adverse impact to living quality. The dosage is based on published clinical studies.
  Other Names: SBRT
  Arms: Camrelizumab Plus Stereotactic Body Radiotherapy

SUMMARY:
We intend to compare the efficacy and safety of immunotherapy plus stereotactic body radiotherapy at oligometastatic lesions and immunotherapy alone among patients with oligometastatic nasopharyngeal carcinoma whose primary lesion has been well controlled after radical local-regional treatment through this multicenter randomized phase 3 trial.

DETAILED DESCRIPTION:
We intend to apply camrelizumab plus stereotactic body radiotherapy at oligometastatic lesions to patients with oligometastatic nasopharyngeal carcinoma whose primary lesion has been well controlled after radical treatment through this multicenter randomized phase 3 trial to investigate whether stereotactic body radiotherapy at oligometastatic lesions on the basis of immunotherapy can achieve clinical cure among a part of patients with distant metastasis and improve their overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; 18-70 years of age.
2. Primary lesion and regional lymph nodes completed radical radiotherapy 3 months before stereotactic body radiotherapy and diseases well controlled.
3. Underwent at least first-line systemic chemotherapy, regardless of regimen and curative effect.
4. Imageological evidence for oligometastatic lesions (metastatic tissue biopsy preferred but not necessary). The number of total metastatic lesions no more than 5 and the number of metastatic lesions within a single organ no more than 3.
5. ECOG performance status of 0 or 1.
6. Stereotactic body radiotherapy applicable for all metastatic lesions according to MDT.
7. If metastatic lesions have received local treatment (surgery, radiofrequency ablation, radiotherapy etc.):

   * Eligible if treated lesion is well controlled according to imageological examinations, and the lesion does not need stereotactic body radiotherapy.
   * If treated lesion is not controlled according to imageological examinations:

     * Eligible if the treatment is surgery and that stereotactic body radiotherapy is applicable for the treated lesion.
     * Ineligible if the treatment is radiofrequency ablation or radiotherapy.
8. Maximum diameter of brain metastatic lesion no more than 3cm.
9. Maximum diameter of metastatic lesion (brain excluded) no more than 5cm.

   * Maximum diameter of bone metastatic lesion no more than 6cm if attending doctor decides it is safe to apply the treatment.
10. Life expectancy more than 12 weeks.

Exclusion Criteria:

1. Immunotherapy (PD-1/PD-L1 or CTLA-4 monoclonal antibody) failure.
2. CHD no less than grade 2, arrhythmia (QTc interval over 450ms for male and 470ms for female) or cardiac insufficiency.
3. History of severe hypersensitivity to any ingredient of PD-1/PD-L1 or other monoclonal antibody.
4. chemotherapy (cytotoxic or molecular targeted) within 4 weeks before stereotactic body radiotherapy.
5. Imageological evidence for spinal cord compression, or tumor less than 3mm away from spinal cord.
6. Patient with brain metastasis who needs decompression surgery.
7. Other malignancy or malignant hydrothorax.
8. Concurrent known or suspicious autoimmune disease, including dementia and epilepsy.
9. Use of large dose corticosteroids within 4 weeks before study drug administration.
10. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids.
11. Active tuberculosis (TB), anti-TB treatment is ongoing or within 1 year prior to screening
12. Subjects with any active autoimmune disease or history of autoimmune disease, or history of syndrome that requires systemic steroids or immunosuppressive medications, including but not limited to the following: rheumatoid arthritis, pneumonitis, colitis (inflammatory bowel disease), hepatitis, hypophysitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy.
13. Has a known history of human immunodeficiency virus (HIV), has hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
14. Received any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to enrollment.
15. Pregnancy or lactation.
16. Other ineligible patients according to attending doctor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | 2 years
  Progression-free survival is calculated from the date of randomization to the date of death of any cause or the first progress at any site, censored on the last date of tumor evaluation if no progress has happened.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Objective response rate is the rate of patients achieving complete response or partial response for a certain period of time after intervention.
Disease control rate (DCR) | 2 years
  Disease control rate is the rate of patients achieving complete response, partial response or stable disease for at least 4 weeks after intervention.
Clinical benefit rate (CBR) | 2 years
  Clinical benefit rate is the rate of patients achieving complete response, partial response or stable disease for at least 6 months after intervention.
Median overall survival (OS) | 2 years
  Overall survival is calculated from the date of randomization to the date of death of any cause, censored on the last date of known survival if no death has happened.
Adverse events | 2 year
  NCI-CTC5.0 and RTOG standards are adopted, and acute subjective toxicity, acute objective toxicity and late subjective toxicity are included.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 2 years.
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China